CLINICAL TRIAL: NCT00491998
Title: Randomised, Double-blind, Double-dummy, Two-period, Cross-over Study to Determine the PK, PD and Safety of Multiple Doses of V1512 Effervescent Tablets in Parkinson's Disease Patients Compared to Sinemet® Oral Tablets
Brief Title: PK, PD and Safety of Multiple Doses of V1512 Tablets in PD Patients Compared to Standard Levodopa/Carbidopa Oral Tablets
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vernalis (R&D) Ltd (Industry)
Collaborators: Cita NeuroPharmaceuticals (Industry); Syneos Health (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: V1512-2PD01
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — entacapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2-hourly dosing (Experimental): 6 Doses of IMP at 2-hourly intervals
  Interventions: Drug: V1512
- 3-hourly dosing (Experimental): 4 doses of IMP at 3-hourly intervals
  Interventions: Drug: V1512
- 3-hourly dosing plus Entacapone (Active Comparator): 4 doses of IMP plus Entacapone at 3-hourly intervals
  Interventions: Drug: V1512 and Entacapone

INTERVENTIONS:
Drug: V1512 — 6 doses of IMP at 2-hourly intervals
  Arms: 2-hourly dosing
Drug: V1512 — 3-hourly dosing
  Arms: 3-hourly dosing
Drug: V1512 and Entacapone — 4 doses of IMP and Entacapone at 3-hourly intervals
  Arms: 3-hourly dosing plus Entacapone

SUMMARY:
The purpose of the study is to determine if the pharmacokinetic profile of V1512 is similar or better than existing medications for the treatment of Parkinson's Disease

DETAILED DESCRIPTION:
The pharmacokinetics of V1512 effervescent tablet has been evaluated in healthy volunteers, however not fully in PD patients. This study aims to evaluate the PK profiles in PD patients of different dosing schedules of V1512 effervescent tablet compared to the profiles after standard L-dopa/carbidopa (Sinemet) over the course of the day. Two dosing schedules have been chosen to evaluate a possible relation between dosing interval and 'ON' time, with and without associated dyskinesia. Similar dosing schedules with the comparator Sinemet are commonly employed in the treatment of fluctuating PD patients. Patients assigned to cohort 3 will also take a dose of entacapone concomitantly with each dose of V1512 or Sinemet, thereby allowing the kinetics and dynamics of.V1512 and Sinemet to be compared in the presence of COMT inhibition.

Safety and tolerability of the dosing regimens in patients will also be assessed further in this double-blind study

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, >30 years of age of any race;
2. A Body Mass Index between 18.5 and 29.9 kg/m2 (inclusive);
3. Clinical diagnosis according to the Brain Bank diagnostic criteria of idiopathic Parkinson's Disease (2 of 3 cardinal symptoms - bradykinesia, rigidity, tremor -must be present, with a positive response to L-dopa);
4. Presence of fluctuations in motor performance with >2 hours inclusive of daytime OFF episodes (not applicable for cohort 1 patients);
5. At least 1 hour delay to ON time with afternoon doses;
6. Discontinued use of COMT inhibitors (cathecol-o-methyl transferase) for at least 2 weeks prior to study entry (not applicable for cohort 3 patients);
7. Stable doses of dopamine agonists or selegiline for at least 2 weeks before entry into the study;
8. Stable comorbidity for 4 weeks;
9. Female patients must be of non-childbearing potential (post-menopausal or physically incapable of childbearing);
10. Willing and able to give informed consent according to national legal requirements prior to initiation of any study-related procedures

Exclusion Criteria:

1. Clinically relevant abnormal vital sign values or safety laboratory data.
2. Patients who smoke and are unable to refrain from smoking during the in-clinic period
3. Diagnosis of atypical parkinsonism;
4. A history and/or the presence of gastro-intestinal disorders (or surgery) that could interfere with absorption of the test medication;
5. A history of intolerance or clinically relevant allergy to L-dopa and/or carbidopa taken in any formulation or combination;
6. A history of intolerance or clinically relevant allergy to entacapone or any ingredients of Comtan (cohort 3 patients only)
7. Any other condition which, in the opinion of the Investigator, would interfere with optimal participation in the study e.g. inability to complete patient diary;
8. Participation in any clinical study or receiving treatment with another investigational drug within 30 days or 5 half lives (whichever is longer) before the screening visit;
9. Blood donation within 3 months before study participation;
10. History of neuroleptic malignant syndrome (NMS) or NMS-like syndromes, or non-traumatic rhabdomyolysis;
11. Patients taking non-selective MAO inhibitors;
12. Patients with a history of, or clinical indication of, narrow angle glaucoma;
13. Patients with a history of, or clinical indication of, malignant melanoma;
14. Patients with a history of, or clinical indication of, depression or psychosis;
15. Patients taking iron containing medications (ferrous sulphate, ferrous gluconate)

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2006-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
to characterise the plasma concentrations of L-dopa after repeated doses of V1512 in fluctuating PD patients compared to standard L-dopa/carbidopa (Sinemet) over the course of the day | 4 weeks

SECONDARY OUTCOMES:
correlate plasma concentrations with response to therapy; | 4 weeks
further characterise the safety and tolerability profile for each treatment | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fabrizio Stocchi, MD, PhD, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele Pisana, Roma, Rome, Italy

REFERENCES:
- [Derived] Stocchi F, Vacca L, Grassini P, Pawsey S, Whale H, Marconi S, Torti M. L-Dopa Pharmacokinetic Profile with Effervescent Melevodopa/Carbidopa versus Standard-Release Levodopa/Carbidopa Tablets in Parkinson's Disease: A Randomised Study. Parkinsons Dis. 2015;2015:369465. doi: 10.1155/2015/369465. Epub 2015 Jun 10. PMID 26171276